CLINICAL TRIAL: NCT01080092
Title: Effect of Stress-management and Biofeedback on Craving in Smoking Abstinence: A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/020
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Smoking Cessation
Keywords: smokers
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- breathing technique group (Experimental): technique as a stress management technique, reinforced by biofeedback
  Interventions: Behavioral: breathing technique
- no breathing technique (Placebo Comparator): the control group reads a paper on the properties and components of tobacco and on behavioural strategies to cope with craving
  Interventions: Behavioral: behavioral strategies

INTERVENTIONS:
Behavioral: breathing technique — breathing technique as a stress management technique, reinforced by biofeedback
  Arms: breathing technique group
Behavioral: behavioral strategies — the control group reads a paper on the properties and components of tobacco and on behavioural strategies to cope with craving
  Arms: no breathing technique

SUMMARY:
Craving is one of the most prominent reasons for relapse after smoking cessation. Mainly pharmacological aids (NRT, bupropion, varenicline) try to counter this condition. This project aims to evaluate the effect of stress-management and a short breathing technique, reinforced by means of visualisation , on the experience of craving in smokers who are prepared to stay abstinent for at least 3 hours before the start of the intervention. It is expected that this strategy can provide supplementary gains in craving control.

ELIGIBILITY:
Inclusion Criteria:

* smokers (at least 10 cigarettes/day);
* 18 years of age or older;
* prepared to stay abstinent for 3 hours before the start of the session;
* not prepared to stop smoking;
* Dutch speaking.

Exclusion Criteria:

* acute health related problems;
* psychiatric co-morbidities;
* quit attempts in the past 3 months;
* participation in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Craving at the end of each of two (learning) sessions; | 1 day
  Measurement by means of participant's estimation of feelings of smoking urge and smoking craving (by means of the Minnesota Nicotine Withdrawal Scale) before and immeadiately after each of two intervention sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Hedwig Boudrez, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of University Hospital Ghent — http://www.uzgent.be